CLINICAL TRIAL: NCT04989153
Title: China Health Promotion Foundation/the Second Affiliated Hospital of Zhejiang University, School of Medicine
Brief Title: Nasal Endoscopic Screening and Risk Assessment for Early Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jilin City People's Hospital (Unknown); No. 924 Hospital of the People's Liberation Army of China (Unknown); Kunshan Hospital of Traditional Chinese Medicine (Unknown); Chinese PLA General Hospital (Other); Sichuan Provincial People's Hospital (Other); Affiliated Hospital of Southwest Medical University (Other); Zhongshan Hospital Xiamen University (Other); Jingzhou Hospital of Traditional Chinese Medicine (Unknown); Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 研2015-079
Record Dates: First submitted 2021-07-08; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer; Precancerous Lesion; Helicobacter Pylori Infection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-atrophic gastritis: No atrophic gastritis, The OLGA-0 group;OLGA :Operative Link on Gastritis Assessment)
- mild-moderate atrophic gastritis: The OLGA I-II group;OLGA :Operative Link on Gastritis Assessment)
- severe atrophic gastritis: The OLGA III-IV group;OLGA :Operative Link on Gastritis Assessment)
  Interventions: Diagnostic Test: pepsinogen
- gastric cancer: gastric cancer
  Interventions: Diagnostic Test: pepsinogen

INTERVENTIONS:
Diagnostic Test: pepsinogen — serum pepsinogen diagnosed gastric cancer and precanceous lesion
  Groups: gastric cancer; severe atrophic gastritis

SUMMARY:
Pepsinogens (PGs) can be used for gastric cancer (GC) screening, but the cutoff levels vary among studies, and PG levels are influenced by numerous factors. To examine the diagnostic value of PG levels and Helicobacter pylori (Hp) status for GC and precancerous lesions screening in asymptomatic individuals undergoing health checkup in China.

DETAILED DESCRIPTION:
Pepsinogens (PGs) can be used for gastric cancer (GC) screening, but the cutoff levels vary among studies, and PG levels are influenced by numerous factors. To examine the diagnostic value of PG levels and Helicobacter pylori (Hp) status for GC and precancerous lesions screening in asymptomatic individuals undergoing health checkup in China. We operated a multicenter cross-sectional study of subjects who underwent health checkup at nine International Healthcare Centers in China. All participants underwent gastroscopy and pathological examination, serum PG, 13C-urea breath test, and/or Hp serological current infection marker rapid test, all on the same day. PG related parameters were analyzed in different Hp subgroups and regions.

ELIGIBILITY:
Inclusion Criteria:

intention to undergo gastroscopy during health checkup examination 25-75 years of age.

Exclusion Criteria:

a history of gastric ulcer, gastric polyp, or GC a history of gastrectomy treatment with a proton pump inhibitor in the last month contraindications to gastroscopy a history of Hp eradication a history of abdominal pain, abdominal distention, belching, acid reflux, nausea and other digestive tract symptoms within 1 month incomplete data.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive subjects who underwent regular health checkup at nine International Healthcare Centers in different regions of China
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-03-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
serum pepsinogen levels for GC and precancerous lesions | 1 year
  cutoff values of pepsinogen level for GC and precancerous lesions in different regions in China and in different HP status
Risk factors for GC | 1 year
  the risk factors for GC, according to the logistic regression model

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhao, Master, Principal Investigator — 2nd affiliated hospital of Zhejiang university, school of medicine
Locations (9):
- China (9):
  - Jilin City People's Hospital, Jilin, Jilin
  - Chinese PLA General Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Hospital affiliated to AMU (Southwest Hospital), Chongqing
  - No. 924 Hospital of the People's Liberation Army of China, Guilin
  - Jingzhou Hospital of Traditional Chinese Medicine, Jingzhou
  - Kunshan Hospital of Traditional Chinese Medicine, Kunshan
  - Shanghai Changhai Hospital, Shanghai
  - Zhongshan Hospital affiliated to Xiamen University, Xiamen